CLINICAL TRIAL: NCT07135739
Title: Effect of Functional Electrical Stimulation With Mirror Therapy on Upper Limb Functions and Quality of Life in Hemiplegic Children
Brief Title: Functional Electrical Stimulation With Mirror Therapy on Upper Limb Functions and Quality of Life in Hemiplegic Children
Acronym: FESMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabab Mustafa Abdo (Other)
Responsible Party: Sponsor-Investigator, Rabab Mustafa Abdo, Senior physical therapist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005699
Record Dates: First submitted 2025-07-06; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Upper Limb Paresis; Spastic Hemiplegia
Keywords: hemiplegic cerebral palsy; functional electrical stimulation; mirror therapy
MeSH Terms: conditions — Paresis; Hemiplegia | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: They will be randomly assigned into two groups, control group (A) will receive physical therapy program and study group(B) will receive same physical therapy program as control group (A) in addition FES combined with mirror therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) (Active Comparator): control group (A) will receive physical therapy program The exercise session for one hour for each child in both groups, conducted 3times/ week for 3 successive months.
  1. Flexibility exercises for shorted muscles and spastic muscles.
  2. Strengthening training focusing on the trunk lower limb and upper limb muscles for weak muscles.
  3. Postural control exercise in different positions and different surfaces
  4. General endurance training (Sherief et al., 2020).
  5. Exercises to facilitate hand function including basic reaching grasping, carrying, release and the more complex skills of in-hand manipulation and bilateral hand use were conducted.
  Interventions: Other: Physical therapy program
- Group (B) (Experimental): Group (B) will receive the same physical therapy program as group (A) in addition to combined FES (wrist extensors) and mirror therapy while doing specific exercises (including, grasping and release) conducted 3 times / week for 3 successive months.
  1. The treatment will be explained to every child and his/her parent emphasizing its benefits.
  2. Subjects were treated with a combination therapy of task specific mirror therapy and functional electrical stimulation, consisting of two tasks, for a total duration of thirty minutes.
  3. The subject was positioned on a height adjustable table with the mirror placed in front of the midline.
  4. The positive electrode and negative electrode of the muscle stimulator were placed over the muscle belly of the wrist extensors on forearm over the motor point of extensor digitorum communis/ extensor carpi radialis brevis/ extensor carpi radialis longus (between one-third and half-way from the proximal end of the dorsal forearm) of the affected upp
  Interventions: Device: funcional Electrical stimulation combined with mirror therapy; Other: Physical therapy program

INTERVENTIONS:
Device: funcional Electrical stimulation combined with mirror therapy — * Subjects were treated with a combination therapy of task specific mirror therapy and functional electrical stimulation, consisting of two tasks, for a total duration of thirty minutes.
  * The subject was positioned on a height adjustable table with the mirror placed in front of the mid line.
  * The positive electrode and negative electrode of the muscle simulator were placed over the muscle belly of the wrist extensors on forearm over the motor (between one-third and half-way from the proximal end of the dorsal forearm) of the affected upper limb.
  * The subject was then instructed to observe the mirror reflection for one to two minutes, trying to visualize the mirror image as the affected limb, asked to perform slow, easy to achieve simultaneous bilateral movements (perceived bilateral movements) while continuing to look at ,with the affected limb performing synchronously with the duty cycle of electrical stimulation.
  Arms: Group (B)
Other: Physical therapy program — The program will be applied to all children in both groups (A and B). The exercise session for one hour for each child in both groups, conducted 3times/ week for 3 successive months.
  1. Flexibility exercises for shorted muscles and spastic muscles.
  2. Strengthening training focusing on the trunk lower limb and upper limb muscles for weak muscles.
  3. Postural control exercise in different positions and different surfaces
  4. General endurance training (Sherief et al., 2020).
  5. Exercises to facilitate hand function including basic reaching grasping, carrying, release and the more complex skills of in-hand manipulation and bilateral hand use were conducted.

SUMMARY:
The goal of this clinical trial is to To investigate the combined effect of functional electrical stimulation and mirror therapy on:Quality of life and UL function in children with hemiplegia,Their age will be ranged from 5 to 10 years. The main question[s] it aims to answer [is/are]:Does the combination of functional electrical stimulation and mirror therapy have effects on upper limb function and Quality of life in children with hemiplegia? They will be randomly assigned into two groups, control group (A) will receive physical therapy program and study group(B) will receive same physical therapy program as control group (A) in addition FES combined with mirror therapy.

DETAILED DESCRIPTION:
The program will be applied to all children in both groups (A and B). The exercise session for one hour for each child in both groups, conducted 3times/ week for 3 successive months.

1. Flexibility exercises for shorted muscles and spastic muscles.
2. Strengthening training focusing on the trunk lower limb and upper limb muscles for weak muscles.
3. Postural control exercise in different positions and different surfaces
4. General endurance training .
5. Exercises to facilitate hand function including basic reaching grasping, carrying, release and the more complex skills of in-hand manipulation and bilateral hand use were conducted.

Group (B) will receive the same physical therapy program as group (A) in addition to combined FES (wrist extensors) and mirror therapy while doing specific exercises (including, grasping and release) conducted 3 times / week for 3 successive months.

1. The treatment will be explained to every child and his/her parent emphasizing its benefits.
2. Subjects were treated with a combination therapy of task specific mirror therapy and functional electrical stimulation, consisting of two tasks, for a total duration of thirty minutes.
3. The subject was positioned on a height adjustable table with the mirror placed in front of the midline.
4. The positive electrode and negative electrode of the muscle stimulator were placed over the muscle belly of the wrist extensors on forearm over the motor point of extensor digitorum communis/ extensor carpi radialis brevis/ extensor carpi radialis longus (between one-third and half-way from the proximal end of the dorsal forearm) of the affected upper limb.
5. The subject was then instructed to observe the mirror reflection for one to two minutes, trying to visualize the mirror image as the affected limb.
6. Once the subject got engaged with the mirrored limb they were asked to perform slow, easy to achieve simultaneous bilateral movements (perceived bilateral movements) while continuing to look at the reflected image, with the affected limb performing synchronously with the duty cycle of electrical stimulation.
7. The exercises that performed were active wrist extension and fingers extension in mid-prone and pronated forearm, task specific grasping and releasing of a half-litre bottlereleasing cube and placing cubes. Exercises to facilitate hand function including basic reaching, grasping, carrying, release) if the patient could produce an activity in the muscles above the threshold, music broadcasts from the machine.
8. The other half an hour of the session the child will do the rest of exercises described for group (A).

ELIGIBILITY:
Inclusion Criteria:

* Their age will range from 5 to 10 years.
* Spasticity grade range from 1+ to 2, according to Modified Ashworth Scale (
* They will be able to follow instructions.

Exclusion Criteria:

Children will be excluded if they have any of the following criteria:

* Loss of sensation
* The presence of visual impairments.
* Musculoskeletal problems or fixed deformities in the upper extremities.
* Seizures.
* Surgical interference in upper limbs.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male and female
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
functional ability | 3 successive months.
  functional ability is assesed by The Pediatric Evaluation of Disability Inventory (PEDI) is an interview-based tool that assesses functional abilities, level of independence and extent of modification needed for a child to carry out functional activities. Originally published in 1992 by Haley et al., it has been translated into multiple languages and developed into a computer-adaptive test called Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT).
  It is scored on a four-point scale:
  0 - unable to perform the task
  1. - can perform the task with assistance
  2. - can perform the task independently but with some difficulty
  3. - can perform the task independently and without difficulty
Quality of Life(Qol) | 3 months
  Quality of life will be assessed by The Pediatric Quality of Life Inventory (PedsQL
  The PedsQL 4.0 Generic Core Scales instrument is the last version of PedsQL contain 23-items, including formats for typically developing children and adolescents 2 to 18 years old, and consists of the following:
  Physical functioning (8 items). Emotional functioning (5 items). Social functioning (5 items). School functioning (5 items).
  Each item of the instrument is scored on a 5-point scale from 0- 4 for ages 8-18, (0 = never a problem, 1 = almost never a problem, 2 = sometimes a problem, 3 = often a problem, 4 = almost always a problem) ad 3-point scale for young child self-reporting (ages 5- 7) as following (0 = not at all a problem, 2 = sometimes a problem, 4 = a lot of a problem) the large score means worst symptoms , scores are linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) in which high score means better condition.
Range of motion | 3 months
  A goniometer will be used to evaluate active range of motion of wrist extension. The child will sit on chair and the examiner palpates the relevant bony landmarks and aligns the goniometer and the child moves the joint through the available range of motion.
  , the ROM will be measured as follow: Wristn extension: Centre the fulcrum of the goniometer over the lateral aspect of the wrist over the triquetrum and align the stabilized arm with the lateral midline of the ulna using the olecranon process and ulna styloid for reference. Align the moving arm of the goniometer with the lateral midline of the fifth metacarpal.
hand grip strength | 3 months
  Children will sit on chair with neutral shoulder adduction and rotation, 90° flexion of the elbow, forearm and wrist in neutral on arm rest and ask to carry out the movement with maximum strength while the examiner held the device. During the assessment of strength, all the children will advise to grip the dynamometer with thumb facing the fingers and fingers alongside each other and try to do their effort to assess hand grip strength
hand function | 3 months
  The Quality of Upper Extremity Skills Test (QUEST) is an outcome measure designed to evaluate movement patterns and hand function in children with CP. The QUEST is both reliable and valid. The QUEST was developed specifically for children with spastic CP in order to provide one of several outcome measures for a clinical trial on upper limb casting

IPD SHARING:
Plan to Share IPD: No